CLINICAL TRIAL: NCT03960164
Title: Safety Use of Photosynthetic Dermal Scaffolds for the Treatment of Acute Wounds
Brief Title: Dermal Regeneration Photosynthetic Matrix
Acronym: HULK
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Hospital del Salvador (Other); SymbiOx Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SymbiOx
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2022-07

CONDITIONS: Skin Wound
Keywords: Acute skin lesion; Chronic skin ulcer; Traumatic skin lesion; Photosynthetic matrix; Photosynthesis induced regeneration; Tissue regeneration

STUDY DESIGN:
Intervention Model Description: Single group to test safety of the treatment
Masking Description: There will be no masking of the treatment for researchers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient group (Experimental): The group of patients included in the study following inclusion criteria with local (wound) and systemic test values prior and after to the application of the DRPM.
  Interventions: Combination Product: Dermal regeneration photosynthetic matrix (DRPM)

INTERVENTIONS:
Combination Product: Dermal regeneration photosynthetic matrix (DRPM) — Primary Procedure: DRPM implantation
  1. Wound bed preparation and cleaning.
  2. DRPM implantation.
  3. Illumination with LED device.
  Secondary Procedure: Autologous partial skin graft

SUMMARY:
The aim of the study is to demonstrate that dermal regeneration photosynthetic matrix applied in patients with acute clean skin wound is safe.

DETAILED DESCRIPTION:
Safety of the dermal regeneration photosynthetic matrix (DRPM) will be conducted at: 1) Department of Plastic Surgery of Hospital del Salvador, 2) Red UC Christus, and/or 3) Instituto de Neurocirugía (INCA). This safety assessment represents the first objective of this trial, and will be performed in 20 human patients (between 18-65 years old) presenting non-infected acute wounds (confirmed by negative quantitative culture of tissue sample) and homogenous granulation bed. All patients involved in this study will participate only previous approval of the informed consent for the study protocol which has been already accepted by the Research Ethics Committee of the Metropolitan Health Service (approval number: CECSSMO080820018) and each of the affiliated hospitals.

The inclusion criteria of the patients consist of full-thickness skin wounds, homogeneous granulation tissue and negative bacterial count according to quantitative tissue culture. Exclusion criteria will be based on ages under 18 years or over 65 years. Also, patients with autoimmune diseases or immunosuppression will be excluded from the study. Patients with psychiatric disorders that impede decision-making and continue treatment will also be excluded from the treatment, as well as patients with injuries in the face.

Treatment will be performed in two surgical procedures. In the first one, DRPM will be implanted and illuminated with a LED array. Once the photosynthetic scaffold is properly adhered to the wound bed (approximately 21 days), a second surgical procedure will be carried out, where an autologous partial skin graft will be performed on top of the scaffold. In case of a major complication (uncontrollable pain, sepsis, shock), or at the request of the patient, the DRPM will be removed immediately and the standard treatment will be performed for that type of wound. All patients included in the study will be evaluated for local and systemic immune response against DRPM.

Systemic response will be studied by means of hematological, coagulation and biochemical profiles as well as by quantification of plasma cytokines and immune cells in peripheral blood. Hematological profiles will include hematocrit, erythrocytes, hemoglobin, platelets and leukocytes counts, performed by certified clinical laboratory methods. Coagulation tests will include international normalized ratio (INR), prothrombin time (PT) and partial thromboplastin time (PTT). Biochemical profiles will include quantification of blood glucose, creatinine, bilirubin direct and total levels, serum glutamic-oxaloacetic transaminase (SGOT), serum glutamic-pyruvic transaminase (SGPT), alkaline phosphatase and C-reactive protein, as well as clinically relevant enzymatic activities and plasmatic electrolytes (sodium, potassium and chloride). Concentration of inflammatory plasma cytokines (TNF-α, IL-1β, IL-6, IL-8, IL-12p70 and IL-10), as well as the following circulating immune cells: T-cells (CD3+), T-helper cells (CD3+CD4+), cytotoxic T-cells (CD3+CD8+) and their ratio (CD4+/CD8+), B-cells (CD19+) and NK cells (CD16+CD56+) will be quantified. All parameters will be quantified before DRPM implantation (day 0), short-term after implantation (1-3 days), 1 week after implantation and right before autograft procedure. Parameters will be also quantified short-term after autograft (1-3 days), 1 week after autograft and 2 months after autograft.

Additionally, in order to study the local response of DRPM implantation, a biopsy punch will be obtained before (day 0) and 1 week after scaffold implantation, as well as before and 1 week after autografting, and wound regeneration will be evaluated by quantification of cellularization (nuclear staining), presence of macrophages (CD68) and microorganisms (Giemsa) and neovascularization (CD31).

Finally, a final self-evaluation survey will be completed by all patients, where parameters such as pain, itching, burning, light annoyance, smell and general aspect of the wound will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Full-thickness skin wounds.
* Between 18 and 65 years old
* Non-infected wounds (confirmed by quantitative culture of the tissue sample).
* Homogeneous granulation of wound bed.
* Approval of the informed consent for the study protocol.

Exclusion Criteria:

* Ages under 18 years or older than 65 years.
* Comorbidities such as autoimmune diseases, immunosuppression, coronary heart disease or occlusive arterial disease.
* Chronic drug and/or alcohol abuse.
* Psychiatric disorders that impede decision-making and continue treatment.
* Patients suffering from an acute pathology other than the skin injury.
* Full-thickness skin wounds in face.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Systemic response to the implanted scaffold | 3 months
  Percentage of patients presenting adverse effects, measured by hematological, coagulation and biochemical profiles as well as concentration of plasma cytokines and immune cells in peripheral blood.
Local response to the implanted scaffold | 4-5 weeks
  Percentage of patients presenting adverse effects, measured by: abnormal levels of macrophages, microorganisms in the implanted site and/or non-adherence of the scaffold to the wound bed.

SECONDARY OUTCOMES:
Wound closure | 4-5 weeks
  Percentage of patients with complete wound closure.
Patient self-perception | Up to 10 days
  Average percentage of satisfaction of the following parameters: pain, itch, burn, smell and light annoyance after DRPM implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Egaña, PhD., Principal Investigator — Pontificia Universidad Catolica de Chile; Antonio Eblen-Zajjur, MD., PhD., Study Chair — Pontificia Universidad Catolica de Chile
Locations (3):
- Chile (3):
  - Hospital del Salvador, Santiago, RM
  - Instituto de Neurocirugía (INCA), Santiago
  - Red UC Christus, Santiago

REFERENCES:
- [Result] Obaid ML, Camacho JP, Brenet M, Corrales-Orovio R, Carvajal F, Martorell X, Werner C, Simon V, Varas J, Calderon W, Guzman CD, Bono MR, San Martin S, Eblen-Zajjur A, Egana JT. A First in Human Trial Implanting Microalgae Shows Safety of Photosynthetic Therapy for the Effective Treatment of Full Thickness Skin Wounds. Front Med (Lausanne). 2021 Nov 30;8:772324. doi: 10.3389/fmed.2021.772324. eCollection 2021. PMID 34917636
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fmed.2021.772324/full
- See also: Related Info — https://www.symbiox.org/